CLINICAL TRIAL: NCT00002409
Title: A Phase IIIB, Open-Label, Randomized Study of the Effect of an Education Intervention on Virological Outcomes, Adherence, Immunological Outcome, and Health Outcomes in HIV-Infected Subjects From Under-Represented Populations Treated With Triple Nucleoside Therapy (Combivir, Lamivudine 150 Mg/Zidovudine 300 Mg PO BID Plus Abacavir 300 Mg PO BID) for Twenty-Four Weeks
Brief Title: The Effect of Teaching HIV-Infected Patients About HIV and Treatment
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Glaxo Wellcome (Industry)
Organization: NIH AIDS Clinical Trials Information Service (Industry)
Purpose: Treatment
Other Study IDs: 280B; NZTA 4006
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 1999-06

CONDITIONS: HIV Infections
Keywords: Drug Therapy, Combination; Zidovudine; HIV Protease Inhibitors; Lamivudine; Patient Education; Patient Compliance; Reverse Transcriptase Inhibitors; Anti-HIV Agents; Viral Load; abacavir
MeSH Terms: conditions — HIV Infections; Patient Compliance | interventions — lamivudine, zidovudine drug combination; abacavir

INTERVENTIONS:
Drug: Lamivudine/Zidovudine
Drug: Abacavir sulfate

SUMMARY:
The purpose of this study is to see if an HIV-education course can help under-represented, HIV-infected patients. This study examines the areas of faithfulness to drug regimen, level of HIV in the blood, and health status.

DETAILED DESCRIPTION:
Following initial screening, eligible patients are treated with open-label Combivir plus abacavir for 24 weeks. Patients are randomized to undergo the education intervention, Tools for Health and Empowerment (T.H.E.) course plus counseling, or routine counseling only (control group). Measurements and evaluations for assessment of immunologic effects, adherence, and health outcomes are performed at entry (Day 1) and at Weeks 2, 5, 8, 12, 16, and 24.

ELIGIBILITY:
Inclusion Criteria

Patients must have:

* Documented and confirmed HIV infection.
* Limited or no experience with antiretrovirals.
* CD4+ lymphocyte cell count of 50 cells/mm3 or more 14 days prior to study drug administration.
* HIV-1 plasma RNA above 40 copies/ml and less than 100,000 copies/ml within 14 days prior to study drug administration.
* Ability to read, comprehend, and record information in fifth-grade English.
* Ability to attend the 4 sessions of T.H.E. course on Weeks 1-4.

Exclusion Criteria

Co-existing Condition:

Patients with the following symptoms or conditions are excluded:

* Patients suffering from a serious medical condition such as diabetes, congestive heart failure, cardiomyopathy, or other cardiac dysfunction which would compromise the safety of the patient.
* Malabsorption syndrome or other gastrointestinal dysfunction which may interfere with drug absorption or render the patient unable to take oral medication.
* Acute or chronic active hepatitis.

Concurrent Treatment:

Excluded:

Treatment with foscarnet or other agents with required documented activity against HIV-1 in vitro.

Patients with the following prior conditions are excluded:

* A clinical diagnosis of AIDS, according to the 1993 Centers for Disease Control (CDC) AIDS surveillance definition. (CD4 cell counts below 200 cells/mm3 will not be considered AIDS-defining.)
* History of allergy to any study drug.

Prior Medication:

Excluded:

* History of antiretroviral use. Patients with a history of sequential nucleoside monotherapy will be excluded, as will patients with a total antiretroviral history exceeding 6 months.
* Required treatment with immunomodulating agents, such as systemic corticosteroids, interleukins, vaccines, or interferons, within 4 weeks prior to study entry, or an HIV immunotherapeutic vaccine within 3 months prior to entry. Asthmatic patients using inhaled corticosteroids are eligible for enrollment.

Prior Treatment:

Excluded:

Radiation therapy or cytotoxic chemotherapeutic agents received within 4 weeks prior to entry.

Risk Behavior:

Excluded:

Current alcohol or illicit drug use which may interfere with the ability to comply with dosing schedule and protocol evaluation and assessment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200

CONTACTS AND LOCATIONS:
Overall Officials: K Rawlings, Study Chair
Locations (25):
- United States (25):
  - AIDS Healthcare Foundation, Los Angeles, California
  - Oasis Clinic / King Drew Med Ctr, Los Angeles, California
  - Robert Scott MD, Oakland, California
  - Georgetown Univ Med Ctr, Washington D.C., District of Columbia
  - Whitman Walker Clinic/Elizabeth Taylor Med Ctr, Washington D.C., District of Columbia
  - Univ of Miami School of Medicine, Miami, Florida
  - Specialty Med Care Ctrs of South Florida Inc, Miami, Florida
  - Saint Josephs Comprehensive Research Institute, Tampa, Florida
  - AIDS Research Consortium of Atlanta, Atlanta, Georgia
  - Rush Med College / Dept of Infectious Diseases, Chicago, Illinois
  - Encounter Med Group, Oak Park, Illinois
  - New England Med Ctr / Div of Geo Med & Infect Disease, Boston, Massachusetts
  - Jeffrey Bomser Clinic / NJCR, Newark, New Jersey
  - UMDNJ / Dept of Ob/Gyn, Newark, New Jersey
  - Newark Community Health Ctr, Newark, New Jersey
  - Addiction Research and Treatment Corp, Brooklyn, New York
  - Bentley-Salick Med Practice, New York, New York
  - Holmes Hosp / Univ of Cincinnati Med Ctr, Cincinnati, Ohio
  - Allegheny Univ of the Hlth Sciences / Div of Infect Diseases, Philadelphia, Pennsylvania
  - Carolina Family Care/Denmark Med Ctr / P O Box 278, Denmark, South Carolina
  - Univ of Tennessee, Memphis, Tennessee
  - Univ of Tennessee / Div of Infect Dis / Dept of Med, Memphis, Tennessee
  - Southeast Dallas Health Ctr, Dallas, Texas
  - Therapeutic Concepts, Houston, Texas
  - Santa Rosa Med Ctr / Baptist Med Ctr, San Antonio, Texas